CLINICAL TRIAL: NCT04683341
Title: Safety and Efficacy of Tenofovir Alafenamide for Chronic Hepatitis B Patients With Decompensated Liver Disease
Brief Title: Tenofovir Alafenamide in HBV Related Decompensated Liver
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TAF-Deliver
Record Dates: First submitted 2020-11-12; First posted 2020-12-24 (Actual); Last update posted 2020-12-24 (Actual); Status verified 2020-11

CONDITIONS: HBV
MeSH Terms: interventions — tenofovir alafenamide

STUDY DESIGN:
Intervention Model Description: Approximately 100 adults, cirrhotic or non-cirrhotic (capped at 50), CHB patients with hepatic decompensation, will receive initial treatment (Arm A) with or switch (Arm B) to TAF 25 mg/day for 144 weeks. For Initiation Arm, CHB patients with hepatic decompensation, who are currently not under HBV antiviral treatment will be enrolled. For Switch Arm, CHB patients who are currently with hepatic decompensation and virally suppressed under HBV NUC treatment (HBV DNA < 20 IU/mL) will be enrolled.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Arm A - initial TAF treatment group (Experimental): cirrhotic or non-cirrhotic CHB patients with hepatic decompensation and HBV NUC treatment naïve or experienced (except prior TAF) will receive initial treatment (Arm A) with TAF 25 mg/day.
  Interventions: Drug: Tenofovir Alafenamide Tablets
- Arm B - switch to TAF treatment group (Experimental): cirrhotic or non-cirrhotic CHB patients with hepatic decompensation and currently under HBV NUC treatment (except TAF) with HBV DNA < 20 IU/mL within 6 months prior screening will switch (Arm B) to TAF 25 mg/day
  Interventions: Drug: Tenofovir Alafenamide Tablets

INTERVENTIONS:
Drug: Tenofovir Alafenamide Tablets — Approximately 100 adults, cirrhotic or non-cirrhotic (capped at 50), CHB patients with hepatic decompensation, will receive initial treatment (Arm A) with or switch (Arm B) to TAF 25 mg/day for 144 weeks. For Initiation Arm (Arm A), CHB patients with hepatic decompensation, who are currently not under HBV antiviral treatment will be enrolled. For Switch Arm (Arm B), CHB patients who are currently with hepatic decompensation and virally suppressed under HBV NUC treatment (HBV DNA < 20 IU/mL) will be enrolled.

SUMMARY:
TAF is a new prodrug of tenofovir, specifically designed to achieve higher intracellular active drug concentration allowing for dosing of only 25 mg once daily and thus can potentially lower the already relatively low risk of renal toxicity and bone loss with TDF. However, such renal and bone complications with TDF may become more pronounced in decompensated CHB patients10. In the phase 3 trials11, 12, TAF had demonstrated a compatible antiviral effect (noninferior efficacy), and a higher rate of alanine aminotransferase (ALT) normalization to TDF. TAF also demonstrated an improved renal function and less bone loss compared to TDF. Therefore, TAF was approved as the first line therapy for CHB patients with compensated liver function. The lack of data regarding TAF therapy in decompensated CHB patients raised the concern of safety and efficacy of TAF in this group of patients. A small, single arm Phase 2 switch study (GS-US-320-4035; Study 4035; NCT03180619) which has enrolled 31 subjects with CPT scores ≥7, either at time of screening or by history, who were virally suppressed on TDF and/or other oral antiviral agents is currently underway with favorable safety and efficacy results through 48 weeks.[Lim YS, Lin CY, Heo J, et al. EASL 2020, poster SAT442.] While Gilead Study 4035 will continue through 96 weeks of treatment, additional data in this population are thus needed, particularly in CHB patients who have decompensated liver disease and are not being treated and are viremic. Herein, we conduct the present study and aim to investigate the safety and efficacy of TAF in CHB patients with hepatic decompensation.

ELIGIBILITY:
Inclusion Criteria:

* Male or non-pregnant female, age ≥20 years
* Chronic HBV infection with positive hepatitis B surface antigen (HBsAg) for at least 6 months at screening.
* Hepatic decompensation, defined as Child-Turcotte-Pugh (CTP) score ≥7, or the presence of portal hypertension related complications including ascites, hepatic encephalopathy (<grade 2) at screening.
* HBV NUC treatment naïve or experienced (except prior TAF) for Arm A or currently under HBV NUC treatment (except TAF) with HBV DNA < 20 IU/mL within 6 months prior screening for Arm B.
* Patients with either liver cirrhosis or non-cirrhosis (defined by histology, non-invasive assessments, or imaging/clinical based diagnosis).
* Estimated creatinine clearance ≥30 ml/min (using the Cockcroft-Gault method) at screening. (Note: multiply estimated rate by 0.85 for women).
* Willing and able to provide informed consent
* Able to comply with dosing instructions for study drug administration and able to complete the study schedule of assessments

Exclusion Criteria:

* Pregnant women, women who are breast feeding or who believe they may wish to become pregnant during the course of the study.
* Previous recipient of a solid organ (including liver), or bone marrow transplant.
* Severe or uncontrolled comorbidities determined by the Investigator.
* Currently ≥grade 2 hepatic encephalopathy, currently or history (within 60 days) of variceal bleeding, hepatorenal syndrome, refractory ascites or spontaneous bacterial peritonitis; cytopenia of absolute neutrophil count < 750/mm3, or hemoglobin < 8 g/dL, or platelet <30000/mm3; or MELD score ≥30 at screening.
* Malignancy history including hepatocellular carcinoma, except basal cell skin cancer without recurrence for more than 5 years.
* Acute exacerbation of HBV, defined as an elevation of alanine aminotransferase (ALT) activity to more than 10 times the upper limit of normal and more than twice the baseline value.
* On any of the disallowed concomitant medications listed in the prior and concomitant medications list (pg. 16). Subjects on prohibited medications who are otherwise eligible will need a wash out period of at least 30 days prior to the Screening.
* Males and females of reproductive potential who are unwilling to use "effective" protocol-specified method(s) of contraception during the study.

Ages: 20 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-09-01 (Actual); Primary Completion 2021-01-31 (Estimated); Study Completion 2025-04-01 (Estimated)

PRIMARY OUTCOMES:
Complete virological suppression | week 48
  Proportion of patients treated with TAF who achieve complete virological suppression (HBV DNA < 20 IU/ml) at week 48 of TAF therapy in per-protocol (PP) population.

SECONDARY OUTCOMES:
Rate of adverse events | week 48
  Rate of adverse events including serious adverse events and discontinuation at Week 48
Rate of recovery from hepatic decompensation | week 48, 96, and 144
  Rate of recovery from hepatic decompensation (improvement of CTP score ≥1) at week 48, 96, and 144 of TAF therapy in FAS, modified FAS (mFAS) and PP populations.
Liver transplant-free survival | week 48, 96, and 144
  Liver transplant-free survival at week 48, 96, and 144 of TAF therapy in FAS, mFAS and PP populations.
Rate of virological response | week 96, and 144
  Rate of virological response (HBV DNA < 20 IU/ml) at week 96, and 144 of TAF therapy
Rate of ALT normalization | week 48, 96, and 144
  Rate of ALT normalization by local (<40 U/L), and AASLD (male ≤35, female ≤25 U/L) criteria at week 48, 96, and 144 of TAF therapy in FAS, mFAS and PP populations.
Rate of HBeAg loss/seroconversion, HBsAg loss/seroconversion | week 48, 96, and 144
  Rate of HBeAg loss/seroconversion in baseline HBeAg-seropositive patients, HBsAg loss/seroconversion, and change in HBsAg titer at week 48, 96, and 144 of TAF therapy.
Changes of serum creatinine | week 48, 96, and 144
  Changes of serum creatinine from baseline to week 48, 96, and 144 of TAF in mFAS and PP populations.
Changes of calculated creatinine clearance | week 48, 96, and 144
  Changes of calculated creatinine clearance (Cockcroft-Gault) from baseline to week 48, 96, and 144 of TAF in mFAS and PP populations.
Changes in bone mineral density | week 144
  Changes in bone mineral density from baseline to week 144 of TAF in mFAS and PP populations.
Changes in value of transient elastography | week 144
  Changes in value of transient elastography (Fibroscan, kPa) from baseline to week 144 in mFAS and PP populations.
Changes in body mass index | week 48, 96, and 144
  Changes in body mass index (BMI) from baseline to week 48, 96, and 144 of TAF in mFAS and PP populations.
Changes in blood lipid profile | week 48, 96, and 144
  Changes in fasting blood lipid profiles from baseline to week 48, 96, and 144 of TAF in mFAS and PP populations.
Changes in blood glucose | week 48, 96, and 144
  Changes in fasting blood glucose from baseline to week 48, 96, and 144 of TAF in mFAS and PP populations.

CONTACTS AND LOCATIONS:
Overall Officials: Ming-Lung Yu, Professor, Principal Investigator — Hepatobiliary Division, Kaohsiung Medical University Hospital
Locations (1):
- Kaohsiung Medical University Hospital, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lavanchy D. Hepatitis B virus epidemiology, disease burden, treatment, and current and emerging prevention and control measures. J Viral Hepat. 2004 Mar;11(2):97-107. doi: 10.1046/j.1365-2893.2003.00487.x. PMID 14996343
- [Background] Liaw YF, Chu CM. Hepatitis B virus infection. Lancet. 2009 Feb 14;373(9663):582-92. doi: 10.1016/S0140-6736(09)60207-5. PMID 19217993
- [Background] Sarin SK, Kumar M, Lau GK, Abbas Z, Chan HL, Chen CJ, Chen DS, Chen HL, Chen PJ, Chien RN, Dokmeci AK, Gane E, Hou JL, Jafri W, Jia J, Kim JH, Lai CL, Lee HC, Lim SG, Liu CJ, Locarnini S, Al Mahtab M, Mohamed R, Omata M, Park J, Piratvisuth T, Sharma BC, Sollano J, Wang FS, Wei L, Yuen MF, Zheng SS, Kao JH. Asian-Pacific clinical practice guidelines on the management of hepatitis B: a 2015 update. Hepatol Int. 2016 Jan;10(1):1-98. doi: 10.1007/s12072-015-9675-4. Epub 2015 Nov 13. PMID 26563120
- [Background] European Association for the Study of the Liver. EASL 2017 Clinical Practice Guidelines on the management of hepatitis B virus infection. J Hepatol. 2017 Aug;67(2):370-398. doi: 10.1016/j.jhep.2017.03.021. Epub 2017 Apr 18. PMID 28427875
- [Background] Terrault NA, Lok ASF, McMahon BJ, Chang KM, Hwang JP, Jonas MM, Brown RS Jr, Bzowej NH, Wong JB. Update on Prevention, Diagnosis, and Treatment of Chronic Hepatitis B: AASLD 2018 Hepatitis B Guidance. Clin Liver Dis (Hoboken). 2018 Aug 22;12(1):33-34. doi: 10.1002/cld.728. eCollection 2018 Jul. No abstract available. PMID 30988907
- [Background] Yao FY, Bass NM. Lamivudine treatment in patients with severely decompensated cirrhosis due to replicating hepatitis B infection. J Hepatol. 2000 Aug;33(2):301-7. doi: 10.1016/s0168-8278(00)80371-2. PMID 10952248
- [Background] Fontana RJ, Hann HW, Perrillo RP, Vierling JM, Wright T, Rakela J, Anschuetz G, Davis R, Gardner SD, Brown NA. Determinants of early mortality in patients with decompensated chronic hepatitis B treated with antiviral therapy. Gastroenterology. 2002 Sep;123(3):719-27. doi: 10.1053/gast.2002.35352. PMID 12198698
- [Background] Schiff E, Lai CL, Hadziyannis S, Neuhaus P, Terrault N, Colombo M, Tillmann H, Samuel D, Zeuzem S, Villeneuve JP, Arterburn S, Borroto-Esoda K, Brosgart C, Chuck S; Adefovir Dipivoxil Study 45 Intrnational Investigators Group. Adefovir dipivoxil for wait-listed and post-liver transplantation patients with lamivudine-resistant hepatitis B: final long-term results. Liver Transpl. 2007 Mar;13(3):349-60. doi: 10.1002/lt.20981. PMID 17326221
- [Background] Shim JH, Lee HC, Kim KM, Lim YS, Chung YH, Lee YS, Suh DJ. Efficacy of entecavir in treatment-naive patients with hepatitis B virus-related decompensated cirrhosis. J Hepatol. 2010 Feb;52(2):176-82. doi: 10.1016/j.jhep.2009.11.007. Epub 2009 Dec 16. PMID 20006394
- [Background] Liaw YF, Sheen IS, Lee CM, Akarca US, Papatheodoridis GV, Suet-Hing Wong F, Chang TT, Horban A, Wang C, Kwan P, Buti M, Prieto M, Berg T, Kitrinos K, Peschell K, Mondou E, Frederick D, Rousseau F, Schiff ER. Tenofovir disoproxil fumarate (TDF), emtricitabine/TDF, and entecavir in patients with decompensated chronic hepatitis B liver disease. Hepatology. 2011 Jan;53(1):62-72. doi: 10.1002/hep.23952. Epub 2010 Oct 27. PMID 21254162
- [Background] Chan HL, Fung S, Seto WK, Chuang WL, Chen CY, Kim HJ, Hui AJ, Janssen HL, Chowdhury A, Tsang TY, Mehta R, Gane E, Flaherty JF, Massetto B, Gaggar A, Kitrinos KM, Lin L, Subramanian GM, McHutchison JG, Lim YS, Acharya SK, Agarwal K; GS-US-320-0110 Investigators. Tenofovir alafenamide versus tenofovir disoproxil fumarate for the treatment of HBeAg-positive chronic hepatitis B virus infection: a randomised, double-blind, phase 3, non-inferiority trial. Lancet Gastroenterol Hepatol. 2016 Nov;1(3):185-195. doi: 10.1016/S2468-1253(16)30024-3. Epub 2016 Sep 22. PMID 28404091
- [Background] Buti M, Gane E, Seto WK, Chan HL, Chuang WL, Stepanova T, Hui AJ, Lim YS, Mehta R, Janssen HL, Acharya SK, Flaherty JF, Massetto B, Cathcart AL, Kim K, Gaggar A, Subramanian GM, McHutchison JG, Pan CQ, Brunetto M, Izumi N, Marcellin P; GS-US-320-0108 Investigators. Tenofovir alafenamide versus tenofovir disoproxil fumarate for the treatment of patients with HBeAg-negative chronic hepatitis B virus infection: a randomised, double-blind, phase 3, non-inferiority trial. Lancet Gastroenterol Hepatol. 2016 Nov;1(3):196-206. doi: 10.1016/S2468-1253(16)30107-8. Epub 2016 Sep 22. PMID 28404092
- [Background] Dai CY, Chuang WL, Hou NJ, Lee LP, Hsieh MY, Lin ZY, Chen SC, Huang JF, Hsieh MY, Wang LY, Tsai JF, Wen-Yu, Yu ML. Early mortality in Taiwanese lamivudine-treated patients with chronic hepatitis B-related decompensation: evaluation of the model for end-stage liver disease and index scoring systems as prognostic predictors. Clin Ther. 2006 Dec;28(12):2081-92. doi: 10.1016/j.clinthera.2006.12.016. PMID 17296464